CLINICAL TRIAL: NCT04836416
Title: Appetite Ratings and Eating Patterns
Brief Title: Appetite Variability
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Richard Mattes PhD, RD, Purdue University
Other Study IDs: 2020-1651
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Young Adult/Normal: Age 18-35, BMI 18.5-24.9
  Interventions: Other: Observational
- Young Adult/Overweight and Obese: Age18-35, BMI greater than 25.0
  Interventions: Other: Observational
- Adult/Normal: Age 36-50, BMI 18.5-24.9
  Interventions: Other: Observational
- Adult/Overweight and Obese: Age 36-50, BMI greater than 25.0
  Interventions: Other: Observational
- Older Adult/Nornal: Age 51-65, BMI 18.5-24.9
  Interventions: Other: Observational
- Older Adult/Overweight and Obese: Age 51-65, BMI greater than 25.0
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This study will examine appetitive sensation variability and the relationship between appetitive sensations and energy intake. Investigators believe the methods for assessing and interpretation of appetitive sensations are problematic and mask the true influence of these sensations on eating. This limits the development of guidelines for weight management. To gain a better understanding of the relationship, investigators will track hourly appetite sensations and map these to eating events via time-series analyses to gain new insights on the directionality and magnitude of these relationships. Also, investigators will also examine the association of apetitive ratings with age or gender. This will allow the development of more effective weight management recommendations.

DETAILED DESCRIPTION:
Screening - The study will be advertised through various public media sources (social media, posted flyers, Purdue Today) and a verbal conversation. Participants responding to the advertisements will be scheduled for a screening visit. This meeting will begin with a full description of the study, and investigators will secure informed written consent. Participants will complete questionnaires eliciting demographic (age, biological sex, BMI, fat%), dietary (eating traits), and health (acute and chronic disease history) information. Height and weight will be measured. For those choosing to enroll, investigators will obtain baseline measurements to confirm eligibility. Individuals qualified and volunteering to participate in the trial will complete multiple questionnaires about eating habits ( Meal pattern questionnaire, Power of food scale, 0 Study Materials - Appetite Training Material.pdf 0 Study Materials - ASA24 instruction .pdf 0 Eating Trait questionnaires.pdf 0 Study Materials - Appetite Lexicon Quiz.docx 0 Hourly Appetite and Thirst Ratings.pdf 0 Study Timeline.pdf Emotional eating scale, Eating inventory, Food craving inventory, Adult eating behavior scales, Self-regulation of eating behavior questionnaire, Barrot Impulsiveness scale). Participants will also learn how to record their energy intake through the ASA-24 system. Then, participants will get training on the lexicon of appetite sensations with a video tutorial, followed by an online quiz to confirm their understanding of the concepts. At least 90% of correct responses are required to pass the appetite lexicon training. Failure to satisfactorily convey an understanding of the concepts will result in an offer to repeat the training two more times or be rejected from the study. Study Procedure - Enrolled participants will have a virtual meeting with a researcher (E. Cheon) once a week through Zoom to remind participants about the necessity and method for recording of appetite/thirst ratings, dietary recalls, and physical activity to be completed during three days (2 non-consecutive weekdays and

1 weekend day). Participants will be asked to report to the laboratory for instruction on recording appetitive sensations (hunger, fullness, thirst), food intake, physical activity at baseline (week1), week 9, and 17 on 3 days (2 non-consecutive weekdays and 1 weekend day). Ratings of hunger, fullness, and thirst will be recorded on their cell phones/computers via a web-based Qualtrics survey every waking hour for 3 days. All entries are time and date stamped to ensure the ratings are made at the intended times. Participants will be provided hourly alarms to ensure regular recording.

Concurrently, participants will keep a diet record with an ASA-24 system and free-living energy expenditure will be measured using a physical activity tracking application on the same days of appetite ratings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Body weight fluctuation of <2.5 kg in the past 3 months.

Exclusion Criteria:

1. Having an acute disease.
2. Planning to initiate or terminate medication known to affect appetite.
3. Planning to initiate or terminate lifestyle behaviors that could affect energy balance
4. Age <18 or >65 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Hunger | 4 months
  A positive association between hunger and eating frequency.
Thirst | 4 Months
  A positive association between thirst and energy intake from beverages.
Fullness | 4 Months
  A positive association between fullness and portion size.
Energy Intake | 4 Months
  A positive association between combined hunger (determinant of eating frequency) and fullness (determinant of portion size) ratings and energy intake.
Age | 4 Months
  A negative association between appetitive sensation intensities and age.
Gender | 4 Months
  No significant association between appetitive sensation intensities and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No